CLINICAL TRIAL: NCT04883255
Title: Cannabis Use, Cognition, and the Endocannabinoid System in HIV
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Arpi Minassian, Clinical Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 210323; R01DA051295 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: HIV-1-infection
Keywords: cannabis; HIV; THC; cannabidiol
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HIV-positive subjects (Experimental): Adult human subjects seropositive for HIV-1
  Interventions: Drug: 10 mg Δ9-tetrahydrocannabinol (THC); Drug: 600 mg cannabidiol (CBD); Drug: Placebo
- Healthy Comparison Volunteers (Active Comparator): Adult human subjects without HIV
  Interventions: Drug: 10 mg Δ9-tetrahydrocannabinol (THC); Drug: 600 mg cannabidiol (CBD); Drug: Placebo

INTERVENTIONS:
Drug: 10 mg Δ9-tetrahydrocannabinol (THC) — 5-day course of orally-administered THC (dronabinol), 10 mg
Drug: 600 mg cannabidiol (CBD) — 5-day course of orally-administered CBD, 600 mg
Drug: Placebo — 5-day course of orally-administered placebo

SUMMARY:
Understanding how co-morbidities in persons with HIV (PWH) such as substance use affect risk-taking, decision-making, and other cognitive behaviors is important given implications for everyday functioning and transmission risk. The high prevalence of cannabis use in PWH, medicinally and recreationally, may indicate disease severity, impart therapeutic benefits, or adverse consequences. In fact, cannabis is recommended to those with HIV to alleviate nausea, improve appetite, relieve pain, and lift mood. To-date, the consequences of cannabis use in PWH remain unclear as do potential interactions with HIV treatments. In healthy participants, heavy cannabis use is associated with cognitive deficits e.g., risky decision-making, response disinhibition and inattention, but pro-cognitive effects in PWH may exist at mild use levels due to its anti-inflammatory and anti-excitotoxic properties. Furthermore, little has been done to determine the effects of cannabis use on the endocannabinoid (EC) system in general or in PWH. This study will determine the effects of the two primary cannabis constituents (Δ9-tetrahydrocannabinol [THC], cannabidiol [CBD]) vs. placebo on risky decision-making, response inhibition, reward learning, temporal perception, and motivation, plus EC and homovanillic acid (HVA; a surrogate for dopamine activity) levels in HIV+ and HIV- subjects. Participants with infrequent cannabis use will undergo baseline cognitive testing and biomarker assays with antiretrovirals (ART) use quantified. They will be randomized to a 5-day course of either THC, CBD, or placebo and return for follow-up testing and re-assaying of ECs and HVA levels.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18-65
2. Possess the capacity to provide informed consent to a set of neurobehavioral, neuromedical and cognitive assessment procedures. Individuals unable to provide such consent will not be enrolled into the study.
3. Willing to confirm self-reported HIV using a rapid test: HIV status will be determined using the MedMira Rapid Test (Halifax, Nova Scotia, Canada). If the result differs from the participant's self-report a confirmatory Western Blot will be performed.
4. Willing to abstain from cannabis for at least 1 week prior to the baseline visit and during the study. Although there is no definitive method for determining abstinence over this period, abstinence will be confirmed as best as possible by using an oral fluid testing device (Draeger 5000) employed by law enforcement officers to detect recent cannabis use. An oral fluid value of > 5ng suggests recent use, although in some cases it has been reported that individuals may show > 5ng up to 20 hours after use. Thus, should the oral fluid sample indicate > 5ng THC, the assessment may be canceled and rescheduled.

Exclusion Criteria

* Inability to provide informed consent
* Significant chronic renal disease (unrelated to HIV), significant chronic pulmonary disease (unrelated to HIV), or Hepatitis C Virus infection
* Head injury with loss of consciousness for greater than 30 minutes or resulting in neurologic complications
* Seizure disorder
* Demyelinating diseases or other non-HIV neurological disorders
* Pregnancy
* Acute or recent or previous clinically disabling stroke or previous cerebrovascular events
* Lifetime history of schizophrenia or other psychotic disorders, or bipolar disorder.
* Beck Depression Inventory-II (BDI-II) score is greater than or equal to 29 (severe depression) or suicidal ideas are endorsed on the BDI-II or a Center for Epidemiological Studies-Depression Scale (CES-D) subscale measuring suicidal ideation
* Substance use disorder (mild, moderate or severe) within the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
change in Iowa Gambling Task score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect increased risk-taking
change in Human Temporal Bisection Task score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Scores reflect fast or slow perception of timing.
change in Probabilistic Learning Task score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect poorer learning.
change in Progressive Ratio Task score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect lower motivation or willingness to work for a reward.
change in Continuous Performance Task score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect worse attention.
change in human Behavioral Pattern Monitor activity and exploration score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Higher scores reflect motor hyperactivity and increased exploration.
change in prepulse inhibition percentage score from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower scores reflect worse sensorimotor gating.
change in cerebrospinal fluid (CSF) anandamide (AEA) quantity from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower AEA signifies less amounts of this endocannabinoid in the central nervous system.
change in cerebrospinal fluid (CSF) 2-Arachidonoylglycerol (2-AG) quantity from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower 2-AG signifies less amounts of this endocannabinoid in the central nervous system.
change in cerebrospinal fluid (CSF) homovanillic acid (HVA) quantity from baseline to post-intervention | baseline and 5 days after drug initiation
  This is an experimental measure and not a scale with specific anchor points. Lower HVA signifies less amounts of this dopamine metabolite in the central nervous system.

CONTACTS AND LOCATIONS:
Overall Officials: Arpi Minassian, Ph.D., Principal Investigator — UC San Diego
Locations (1):
- UC San Diego Medical Center-Hillcrest, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No